CLINICAL TRIAL: NCT06837350
Title: Music on Post-cesarean
Brief Title: Effects of Music on Post-Cesarean Pain, Anxiety, Breastfeeding and Mother Infant Attachment Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Principal Investigator, Nuran Nur AYPAR AKBAĞ, Asisstant Professor, Obstetrics and gynecology nursing., Sinop University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024/301
Record Dates: First submitted 2025-01-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Cesarian Section; Bonding; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Control Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- music group (Experimental): music group
  Interventions: Other: Music intervention
- control group (No Intervention): control group

INTERVENTIONS:
Other: Music intervention — Listening to Turkish Music
  Arms: music group

SUMMARY:
The physiological effects of music therapy include creating a behavioral change and changing the mood by reducing psychophysiological stress, pain, anxiety and isolation. Music has the ability to create deep relaxation. It is known to have relieving effects on insomnia. In addition, it has been reported that music therapy application before and during birth reduces labor pain and reduces postpartum anxiety and depression levels. The postpartum period, which begins with the birth of the newborn, covers the 6-8 week period that it takes for the changes that occur in the woman's body during pregnancy to return to its pre-pregnancy state. This period is an important transition period in which physical, social and emotional changes occur in mothers. In addition to rapid anatomical and physiological changes, mothers experience a difficult process in which the transition to motherhood is experienced, new roles and responsibilities are assumed, and relationships with their spouses and other family members are reorganized. Although a woman begins to feel the changes that having a baby creates in her daily life during pregnancy, she usually experiences the biggest change after the baby is born. The period when the first emotional bond between the newborn and her family is formed and a sense of trust develops is defined as mother-baby bonding. Many factors affect mother-baby bonding in the postpartum period, which is the most important time when the bond established between the expectant mother and the baby during pregnancy, referred to as prenatal bonding, is strengthened after birth. It is particularly affected by the mother's upbringing, as well as her experiences during pregnancy, birth, puerperium, and the baby's first months. Healthy and early interaction between mother and baby initiates a healthy bonding process.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being in the third trimester (up to 2 weeks before the planned cesarean delivery date)
* Being primigravida
* Having a single fetus
* Not having a hearing problem
* Voluntarily participating in the study

Exclusion Criteria:

* Having any chronic disease
* Having a risky pregnancy condition (gestational diabetes, gestational hypertension, preeclampsia, etc.)
* Having a psychiatric medical diagnosis and using medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-13 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS)-pain | On the second day after C-section and the end of the 1st week postpartum, change from first pain level an average of 20 minutes.
  Pain Level by Visual Analog Scale The patient marks the pain he/she feels on a scale of 10 cm (100 mm), pain point 1 means "no pain", pain point 10 means "worst pain possible."
Postpartum Specific Anxiety Scale (PSAS) | On the second day after C-section and the end of the 1st week postpartum, change from first pain level an average of 30 minutes.
  Anxiety Level by Postpartum Specific Anxiety Scale (PSAS). The VAS-anxiety is a 10 cm line used to measure perceived anxiety intensity, with endpoints labeled "No Anxiety" and "Worst Anxiety Imaginable." It meansthat those who score 73 and below on the scale have lowpostpartum anxiety levels, and those who score 101 andabove have a high level of anxiety.
Mother and Newborn Information Form I and I | On the second day after C-section and end of the 1st postpartum week
  It will be evaluated with the Mother and Newborn Information Form I and II created by the researchers. Breastfeeding information will be assessed with this form.
Mother Infant Attachment | On the second day after C-section and end of the 1st postpartum week
  It will be evaluated with the Mother-Infant Attachment Scale. The total score ranges from 0 to 24, with higher scores indicating lower mother-infant attachment.

IPD SHARING:
Plan to Share IPD: No
Sharing is not considered appropriate until the article has completed its journal process and is published.